CLINICAL TRIAL: NCT01168362
Title: Evaluation of Coronary Artery Disease With Multidetector-Row Cardiac Computed Tomography in Positive Cardiovascular Risk or Not
Brief Title: Korea Atherosclerosis Study-3
Acronym: KAS3
Status: Completed | Type: Observational
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Soo Lim, Professor, Seoul National University Bundang Hospital
Other Study IDs: M10642140004-06N4214
Record Dates: First submitted 2010-07-22; First posted 2010-07-23 (Estimated); Last update posted 2013-10-25 (Estimated); Status verified 2013-10

CONDITIONS: Cardiovascular Diseases; Cardiovascular Mortality; All-cause Mortality
Keywords: coronary artery disease; cardiovascular risk; pericardial fat
MeSH Terms: conditions — Cardiovascular Diseases; Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Biochemical paramteres including lipid, glucose, insulin, and other novel cardiometabolic factors
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- High risk group: positive cardiovascular risk group
- Low risk group: negative cardiovascular risk group

SUMMARY:
Multidetector-row Computed Tomography (CT) has been introduced for use in the diagnosis of coronary heart disease. The investigators aimed to characterize coronary artery disease in subjects with cardiovascular risk or not, and in particular plaque natures depending on different status of cardiovascular risk. Especially,the investigators will evaluate the relationships between the pericardial fat and severity of stenosis as well as plaque characteristics using logistic regression models.

ELIGIBILITY:
Inclusion Criteria:

* Korean capable of Multidetector-Row Cardiac Computed Tomography (MDCT)

Exclusion Criteria:

* malignancy
* infection
* shock

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: positive cardiovascular risks or not
Sampling Method: Probability Sample
Enrollment: 4000 (Actual)
Dates: Start 2006-02; Primary Completion 2013-03 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Presence of coronary artery disease | 5 years

SECONDARY OUTCOMES:
Mortality | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Soo Lim, MD,PHD, Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam, South Korea